CLINICAL TRIAL: NCT00147316
Title: Japan Alteplase Clinical Trial (J-ACT): Phase 3 Efficacy and Safety Study of Tissue Plasminogen Activator (Alteplase) for Acute Ischemic Stroke Within 3 Hours of Onset
Brief Title: Japan Alteplase Clinical Trial (J-ACT): Efficacy and Safety Study of Tissue Plasminogen Activator (Alteplase) for Ischemic Stroke
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Collaborators: Kyowa Hakko Kogyo Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 527-0110
Record Dates: First submitted 2005-09-05; First posted 2005-09-07 (Estimated); Results first posted 2012-02-24 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Infarction; Brain Ischemia
Keywords: acute stroke; thrombolytic therapy; tissue plasminogen activator
MeSH Terms: conditions — Cerebral Infarction; Brain Ischemia; Stroke | interventions — Tissue Plasminogen Activator

ARMS (1):
- Alteplase (Experimental): 0.6mg/kg intravenous alteplase with 10% being administered as a bolus followed by continuous infusion of the remainder over 1 hour
  Interventions: Drug: Alteplase

INTERVENTIONS:
Drug: Alteplase — 0.6mg/kg intravenous alteplase with 10% being administered as a bolus followed by continuous infusion of the remainder over 1 hour

SUMMARY:
Based on previous studies comparing Duteplase[a recombinant tissue plasminogen activator (rt-PA) very similar to alteplase] doses, we performed a clinical trial with 0.6mg/kg, which is lower than the internationally approved dosage of 0.9mg/kg, aiming to assess the efficacy and safety of alteplase for the Japanese.

DETAILED DESCRIPTION:
Based on previous studies comparing Duteplase ( an rt-PA very similar to alteplase) doses, we performed a clinical trial with 0.6mg/kg, which is lower than the internationally approved dosage of 0.9mg/kg, aiming to assess the efficacy and safety of alteplase for the Japanese.

The primary endpoints were the rate of patients with mRS score of 0-1 at 3 months and the incidence of sICH within 36 hours. Thresholds for these endpoints were determined by calculating 90% confidence intervals of weighted averages derived from published reports. The protocol was defined according to the National Institute of Neurological Disorders and Stroke (NINDS) rt-PA stroke study with slight modifications.

ELIGIBILITY:
Inclusion Criteria:

Patients with acute ischemic stroke within 3 hours of onset, with a clearly defined time of onset

Exclusion Criteria:

1. patients with rapidly improving neurological symptoms or with minor neurological deficit (National Institutes of Health Stroke Scale (NIHSS) score of ≤4) prior to the start of treatment
2. Computed Tomography (CT) evidence of non-minor early ischemic signs (minor early ischemic sign was defined as the involvement of one-third or less of the middle cerebral artery area)
3. CT evidence of cerebral hemorrhage or subarachnoid hemorrhage
4. symptoms suggestive of subarachnoid hemorrhage
5. lactation, pregnancy or suggestive pregnancy; menstruation
6. platelet count below 100,000/mm3
7. heparin administration within 48 hours preceding stroke onset with an elevated activated partial thromboplastin time (APTT); current use of oral anticoagulants with an International Normalized Ratio (INR) of ≥1.7; use of drugs not allowed to be administered concomitantly with alteplase (other thrombolytic agents, ozagrel sodium, argatroban and edaravone) prior to the study treatment
8. major surgery or serious trauma within the preceding 14 days; serious head or spinal cord trauma within the preceding 3 months
9. a history of gastrointestinal or urinary tract hemorrhage within the previous 21 days
10. arterial puncture at a noncompressible site within the preceding 7 days
11. a history of stroke within the preceding 3 months; a history of intracranial hemorrhage or increased risk of intracranial hemorrhage because of cerebral aneurysm, arteriovenous malformation, neoplasm, etc.
12. concurrent severe hepatic or renal dysfunction
13. malignant tumor under treatment
14. a systolic blood pressure of >185 mmHg or diastolic blood pressure of >110 mmHg
15. a need for aggressive treatment to reduce blood pressure to below these limits(14))
16. blood glucose levels of <50 mg/dL or >400 mg/dL
17. acute myocardial infarction(AMI) or endocarditis after AMI
18. concurrent infectious endocarditis, moya-moya disease (Willis circle occlusion syndrome), aortic dissection, neck trauma, etc.; strong suspicion of ischemic cerebrovascular disorder caused by non-thrombotic occlusion or any other hemodynamic condition
19. seizure at the onset of stroke
20. coma (a Japan Coma Scale score of ≥100)
21. an mRS score of ≥2 before stroke onset
22. a history of hypersensitivity to protein preparations
23. difficulty in monitoring for 3 months
24. less than 3 months since any other clinical trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2002-04; Study Completion 2003-09

CONTACTS AND LOCATIONS:
Overall Officials: Takenori Yamaguchi, MD, Study Chair — National Cerebral and Cardiovascular Center, Japan
Locations (1):
- National Cardiovascular Center, Suita, Osaka, Japan

REFERENCES:
- [Result] Yamaguchi T, Mori E, Minematsu K, Nakagawara J, Hashi K, Saito I, Shinohara Y; Japan Alteplase Clinical Trial (J-ACT) Group. Alteplase at 0.6 mg/kg for acute ischemic stroke within 3 hours of onset: Japan Alteplase Clinical Trial (J-ACT). Stroke. 2006 Jul;37(7):1810-5. doi: 10.1161/01.STR.0000227191.01792.e3. Epub 2006 Jun 8. PMID 16763187
- [Derived] Hirano T, Sasaki M, Tomura N, Ito Y, Kobayashi S; Japan Alteplase Clinical Trial Group. Low Alberta stroke program early computed tomography score within 3 hours of onset predicts subsequent symptomatic intracranial hemorrhage in patients treated with 0.6 mg/kg Alteplase. J Stroke Cerebrovasc Dis. 2012 Nov;21(8):898-902. doi: 10.1016/j.jstrokecerebrovasdis.2011.05.018. Epub 2011 Jul 7. PMID 21737309

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alteplase
Started | 103
Completed | 103
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Alteplase
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.9 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 64

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Modified Rankin Scale (mRS) Score of 0-1 at 3 Months
Description: The number of patients with a mRS score of 0-1. The mRS has 6 items, where 0 = No symptoms at all, 1 = No significant disability despite symptoms, 2 = Slight disability, 3 = Moderate disability, 4 = Moderately severe disability, 5 = Severe disability. The higher scores reflect increased disability.
Time Frame: at 3 months
Measure: Number; unit: participants
Arm/Group | Alteplase
Number analyzed (Participants) | 103
participants | 38

2. Primary Outcome: Number of Patients With Symptomatic Intracranial Hemorrhage (sICH) Within 36 Hours
Description: The number of patients with sICH
Time Frame: within 36 hours
Measure: Number; unit: participants
Arm/Group | Alteplase
Number analyzed (Participants) | 103
participants | 6

ADVERSE EVENTS:
Time Frame: 3 Months
Arm/Group | Alteplase
Serious Adverse Events (participants affected / at risk) | 29/103
Other Adverse Events (participants affected / at risk) | 91/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alteplase (N=103)
Acute myocardial infarction (Cardiac disorders) | 1
Asthma aggravated (Respiratory, thoracic and mediastinal disorders) | 1
Atherosclerosis obliterans (Vascular disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Brain herniation (Injury, poisoning and procedural complications) | 1
Brain oedema (Nervous system disorders) | 3
C-reactive protein increased (Investigations) | 1
Cardiac failure NOS (Cardiac disorders) | 1
Carotid artery dissection (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 3
Cerebral infarction (Nervous system disorders) | 7
Depression (Psychiatric disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Haemorrhagic cerebral infarction (Nervous system disorders) | 2
Infection staphylococcal (Infections and infestations) | 1
Intracranial haemorrhage NOS (Nervous system disorders) | 1
Left atrial myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Platelet count decreased (Investigations) | 1
Pneumonia NOS (Infections and infestations) | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Renal failure NOS (Renal and urinary disorders) | 1
Renal impairment NOS (Renal and urinary disorders) | 1
Subdural hygroma (Nervous system disorders) | 1
Tracheal obstruction (Injury, poisoning and procedural complications) | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1
Ventricular arrhythmia NOS (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alteplase (N=103)
Atrial fibrillation (Cardiac disorders) | 7
Ventricular extrasystoles (Cardiac disorders) | 10
Diarrhoea NOS (Gastrointestinal disorders) | 14
Gastrointestinal haemorrhage NOS (Gastrointestinal disorders) | 6
Periproctitis (Gastrointestinal disorders) | 6
Vomiting NOS (Gastrointestinal disorders) | 14
Pyrexia (General disorders) | 15
Hepatic function abnormal NOS (Hepatobiliary disorders) | 7
Pneumonia NOS (Infections and infestations) | 8
Urinary tract infection NOS (Infections and infestations) | 16
Haemorrhagic cerebral infarction (Nervous system disorders) | 37
Headache NOS (Nervous system disorders) | 15
Haematuria (Renal and urinary disorders) | 8
Neurogenic bladder (Renal and urinary disorders) | 7
Hiccups (Respiratory, thoracic and mediastinal disorders) | 6
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 14
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 22
Contusion (Skin and subcutaneous tissue disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other